CLINICAL TRIAL: NCT01150292
Title: Intake of Low Dose of Docosahexaenoic Acid: Effects on Platelet Functions and Redox Status in Diabetic Patients
Brief Title: Effects of Docosahexaenoic Acid (DHA) on Cardiovascular Disease on Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2009.555
Record Dates: First submitted 2010-06-23; First posted 2010-06-24 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2014-02

CONDITIONS: Type 2 Diabetes
Keywords: DHA supplementation; Type 2 diabetic patient; Platelet function
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- DHA - Sunflower oil (Experimental): 400 mg DHA supplementation by day for 2 weeks then placebo for 2 weeks after a wash out period of 6 to 9 weeks
  Interventions: Dietary Supplement: First period DHA
- Sunflower oil - DHA (Experimental): Placebo during 2 weeks then 400 mg DHA supplementation by day for 2 weeks after a wash out period for 6 to 9 weeks
  Interventions: Dietary Supplement: Second period DHA

INTERVENTIONS:
Dietary Supplement: First period DHA — 400 mg DHA supplementation by day for 2 weeks during the first study period
  Arms: DHA - Sunflower oil
Dietary Supplement: Second period DHA — 400 mg DHA supplementation by day for 2 weeks during the second study period
  Arms: Sunflower oil - DHA

SUMMARY:
Aim: to determine the effects of DHA supplementation:

* on the platelet function through their aggregation and the pathway of arachidonic acid metabolism
* on redox status on cells and plasma
* on inflammation in 16 type 2 diabetic patients in a cross-over study comparing DHA (400 mg/day for 2 weeks) vs Sunflower oil (placebo). Each period is separated by a wash-out period of 6 to 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

* woman
* Type 2 diabetes
* Menopausal or aged between 55 and 75 years old
* Recent HbA1c between 6.5-10%
* Oral anti-diabetic drugs or insulin therapy
* Hypertension or antihypertensive drug

Exclusion Criteria:

* Tobacco
* Excessive drinking
* Post-menopausal hormonal treatment
* Treatment by acetylsalicylic acid, clopidogrel, gliclazide, ticlopidine, NSAID
* Secondary cardiovascular prevention
* antioxidant using
* Fish intake >2 times a week
* Anemia <10g/L
* Thrombopenia <110g/L
* Creatinine clearance <30 ml/min and/or proteinuria >1g/L

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Platelet function induced by collagen | 4 blood sampling in 10 to 13 weeks
  4 blood sampling are made during the time of study which expand from 10 weeks (washout period of 6 weeks) to 13 weeks (washout period of 9 weeks):
  * first at the beginning of the first period
  * second at the end of the period (2 weeks after beginning)
  * third at the beginning of the second period
  * fourth at the end of the period (2 weeks after beginning)

SECONDARY OUTCOMES:
Evaluation of cellular and plasmatic redox status | 4 blood sampling in 10 to 13 weeks
  blood sampling are made during the time of study which expand from 10 weeks (washout period of 6 weeks) to 13 weeks (washout period of 9 weeks):
  first at the beginning of the first period second at the end of the period (2 weeks after beginning) third at the beginning of the second period fourth at the end of the period (2 weeks after beginning)

CONTACTS AND LOCATIONS:
Overall Officials: Martine LAVILLE, MD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - Hospices Civils de Lyon, Bron
  - Centre de Recherche en Nutrition Humaine (CRNH) Rhône-Alpes, Pierre-Bénite

REFERENCES:
- [Result] Vericel E, Colas R, Calzada C, Le QH, Feugier N, Cugnet C, Vidal H, Laville M, Moulin P, Lagarde M. Moderate oral supplementation with docosahexaenoic acid improves platelet function and oxidative stress in type 2 diabetic patients. Thromb Haemost. 2015 Aug;114(2):289-96. doi: 10.1160/TH14-12-1003. Epub 2015 Apr 2. PMID 25832443